CLINICAL TRIAL: NCT03814213
Title: Effect of Comprehensive Geriatric Assessment on Short-time Mortality in Elderly
Brief Title: Effect of Comprehensive Geriatric Assessment on Short-time Mortality in Elderly Cancer Patients
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Marianne Ørum, Principal Investigator, University of Aarhus
Other Study IDs: 90-days mortality
Record Dates: First submitted 2019-01-22; First posted 2019-01-23 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Geriatric Assessment; Cancer
Keywords: Comprehensive geriatric assessment; Cancer; Short time mortality
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No-CGA: Patients were not initially offered CGA due to no booking for CGA
- CGA alone: Patients had CGA, but no tailored follow-up upon identified problems
  Interventions: Other: CGA
- CGA with tailored care: CGA and a tailored follow-up and care for 90 days following the CGA
  Interventions: Other: CGA; Other: tailored care

INTERVENTIONS:
Other: CGA — Multi-level Health assessment
  Groups: CGA alone; CGA with tailored care
Other: tailored care — Tailored care based on problems identified by CGA
  Groups: CGA with tailored care

SUMMARY:
Older cancer patients referred to Oncology outpatient Clinic at Aarhus University Hospital have for a period been offered Comprehensive geriatric Assessment (CGA) as part of a routine practice. Oncology Department was responsible for planning the CGA. A number of patients did however not recieve this offer as planning failed. This Group of patients will be compared to patients recieving Geriatric assessment.

Patients recieving CGA is part of a Randomised controlled study (ID: NCT02837679) comparing CGA without 90 days follow-up to CGA with 90 days of Comprehensive geriatric care.

Patients are identified from electronic medical files. Data regarding death is obtained from Medical files.

DETAILED DESCRIPTION:
Inclusion criteria:

* 70 years or more
* Cancer of the head and neck (HNC), lung (LC), upper gastro-intestinal- tract (UGI) or colo-rectal cancer (CRC)
* Referred to the Outpatient Clinic at department of oncology at Aarhus University Hospital for cancer treatment.
* Living in Aarhus, Favrskov, Odder or Skanderborg Municipalities

Exclusion:

- Referred for specialised palliative care

Patients with both newly diagnosed cancer disease and patients with a relapse of previously treated cancer disease are included. Patients qualify for participation regardless of the stage of the cancer disease and regardless if specific cancer treatment is initiated.

The oncology department is responsible for identifying patients and informing of the planned CGA.

All potential patients referred to the oncology outpatient clinic are identified by retrospective review of lists of planned consultations in the oncology department out patient clinic available in the electronic medical file approximately once a week. By this procedure patients who were not informed of the possibility of having a CGA are identified (Group1) Patients who are referred for geriatric evaluation have a complete CGA at baseline. The CGA comprises 7 instruments for assessing health: Activities of Daily Living (ADL) and Instrumental Activities of Daily Living (IADL) for autonomy, Mini Nutritional Status (MNA) for nutritional state, Mini Mental State Examination (MMSE) for Cognitive state, Geriatric Depression Scale 15-item (GDS) for mood and Cumulative Illness Rating Scale - Geriatrics (CIRS-G) for comorbidity and number of daily medication for polypharmacy as previously published. According to CGA, patients were given a CGA-status of "fit", "vulnerable" or "frail". In order to be "fit" all of the following should be present: Independence in ADL and IADL, less than 5 daily medications, no severe comorbidity and no more than 2 well controlled comorbidities, normal cognitive ability and no indications of depression or malnutrition. Information on whether or not the multidisciplinary team initiated any individual action/advice based on the CGA in group 1 and group 2 was registered as well. Interventions initiated by the multidisciplinary team were recorded in four categories: medical changes, nutritional intervention, physical intervention or social intervention. These interventions were registered before randomization was performed Frail and vulnerable patients are offered participation in a controlled randomized study (Clinical trialsID: NCT02837679). Patients are randomly and 1:1 assigned to either: No tailored follow-up (Group 2) or 90 days tailored follow up (group 3). Randomization were performed by REDcap and allocated equally by CGA-status (frail/vulnerable), gender and index tumor site (CRC or no-CRC).

It is not possible to blind patients or the multidisciplinary team of the randomization.

Group 2 has no tailored follow up on the problems found during CGA. Group 3 has 90 days tailored follow-up on problems that were identified during CGA and problems that evolved during the follow-up period.

Tailored follow-up The tailored intervention consists of phone calls, home visits, or contact to community care-takers. A multidisciplinary team consisting of a trained geriatric nurse and a geriatrician specialist performs the follow up. The team can perform clinical investigation of patients, initiate changes in medication, or referral to further investigation. Furthermore transfusion of blood, fluids or i.v. antibiotics could be performed either at home or in the geriatric out patient clinic.

ELIGIBILITY:
Inclusion Criteria:

cancer of head and neck, lung, upper or lower gastro intestinal Canal Referred for evaluation in oncology department out patient Clinic Living in Aarhus, Odder, Favrskov or Skanderborg municipality

-

Exclusion Criteria:

Referred for specialised palliative care

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: older cancer patients referred for oncology out patient Clinic for evaluaation regarding initialisation of treatment All stages of cancer is included, all kind of treatment is accepted including best supportive care.
Sampling Method: Non-Probability Sample
Enrollment: 781 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
short time mortality | 90 days
  dead within 90 days

SECONDARY OUTCOMES:
1 year mortality | 365 days
  dead within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Else M Damsgaard, DMsc, Study Chair — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Geriatric Department Aarhus University Hospital, Aarhus
  - Aarhus University Hospital, Aarhus

IPD SHARING:
Plan to Share IPD: No